CLINICAL TRIAL: NCT07143201
Title: Model Informed Precision Dosing of Oral Ibuprofen for Treatment of Persistent Patent Ductus Arteriosus: A Pilot Randomized Controlled Feasibility Trial
Brief Title: Precision Dosing of Oral Ibuprofen for PDA, A Pilot RCT
Acronym: MIPD-PDA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: McMaster University (Other); Hamilton Academic Health Sciences Organization (Other)
Responsible Party: Principal Investigator, Samira Samiee-Zafarghandy, Principal Investigator, Hamilton Health Sciences Corporation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HiREB #16287
Record Dates: First submitted 2025-08-08; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Patent Ductus Arteriosus; Preterm
Keywords: MIPD-PDA; PDA; Precision Dosing; Ibuprofen
MeSH Terms: conditions — Ductus Arteriosus, Patent; Premature Birth

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The parents of the participants, the professionals performing the echocardiograms and the statistician will be blinded to the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Dosing (Active Comparator): PNA-based standard dosing of ibuprofen [ <= 72 hours PNA: 10/5/5 q24hrs vs >72 hours PNA 20/10/10 q24hrs].
  Interventions: Drug: Standard Dose - Ibuprofen oral suspension
- Precision Dosing (Experimental): PNA-based regimen only for the initial dose, the rest of regimen will be guided by a MIPD, using a Web-Accessible Population Pharmacokinetics Service (WAPPS-PDA).
  Interventions: Drug: Precision Dose - Ibuprofen oral suspension

INTERVENTIONS:
Drug: Standard Dose - Ibuprofen oral suspension — Standard dosing administers ibuprofen without adjustments, starting with an initial loading dose followed by two maintenance doses at 24-hour intervals: 10/5/5 mg/kg for infants aged ≤72 hours, and 20/10/10 mg/kg for those >72 hours old.
  Arms: Standard Dosing
Drug: Precision Dose - Ibuprofen oral suspension — Precision Dosing (Model-Informed Precision Dosing - MIPD): Begins with the same initial loading dose as the Standard Dosing arm, with subsequent doses adjusted based on a Bayesian forecasting model that integrates real-time PK and echocardiographic data.
  Arms: Precision Dosing

SUMMARY:
Newborns born early are at risk for a serious health problem called patent ductus arteriosus (PDA). PDA is a passageway between heart and lung that can cause life-threatening complications such as bleeding in the brain or even death if it remains open and large. When closure of PDA is needed, doctors make every attempt to do it as soon as possible. Ibuprofen is the best drug to close the PDA, but it only works for 50% of small newborns. The investigators have shown before that small newborns handle ibuprofen differently and the amount of active ibuprofen that reaches their blood can be very unpredictable. Studies have shown if enough ibuprofen reaches the body, it can close the PDA. Therefore the investigators designed this study to see whether it is possible to give each newborn the right amount of ibuprofen that their body needs to close the PDA. The investigators will compare two ways to give ibuprofen in a small number of newborns: 1 - standard amount of ibuprofen to everyone, which is the usual care or 2 - ibuprofen doses that will be changed based on how much active ibuprofen has reached the body and how well the newborn's PDA is closing. The investigators will then compare the number of PDAs closed in each group and closely monitor any possible challenges for this new practice. By doing this project, the goals can be summarized as below:

A. Primary goal: To determine if it is feasible to successfully run a larger study in the future.

B. Secondary goals

1. To assess how well and how safely the personalized (MIPD) method works, using a tool called WAPPS-PDA to guide dosing.
2. To compare the effectiveness and safety of the personalized method with standard ibuprofen dosing.
3. To identify drug levels in the blood (Cmin, AUC0-24, AUC0-72) that are associated with complete, partial, or no response to treatment.

DETAILED DESCRIPTION:
Study Design Overview:

This clinical trial is a single-center, pilot, randomized, controlled, triple-blind study designed to evaluate the feasibility and effectiveness of model-informed precision dosing (MIPD) of oral ibuprofen compared to standard dosing for the treatment of Patent Ductus Arteriosus (PDA) in preterm neonates (≤27+6 weeks gestational age). The trial assesses both operational feasibility and clinical outcomes, with a focus on the use of a pharmacokinetic (PK) prediction module provided by the Web-Accessible Population Pharmacokinetics Service-PDA (WAPPS-PDA).

• Standard Dosing Arm: Participants in this arm receive the standard oral ibuprofen regimen used in the unit. Treatment begins with an initial loading dose, followed by two smaller doses administered at 24-hour intervals. While PK samples and targeted echocardiograms are collected at the same intervals as in the precision dosing arm, these data points do not influence dosing decisions.

• Model-Informed Precision Dosing (MIPD) Arm: Participants in this arm initially receive the same loading dose of ibuprofen as those in the standard dosing arm. Subsequent doses are adjusted using real-time PK data and echocardiographic evaluations through the WAPPS-PDA tool. This tool employs a Bayesian forecasting model to analyze blood samples collected at 6, 30, and 54 hours post-initial dose, combining these results with the PDA response level noted in the targeted echocardiograms to dynamically adjust dosing. Dose adjustments are reviewed every 12 hours to ensure tailored treatment based on the neonate's specific pharmacological response, optimizing the chances of effective PDA closure.

ELIGIBILITY:
Inclusion Criteria:

* Neonates with a gestational age of ≤27+6 weeks
* Admitted to the neonatal intensive care unit (NICU) at McMaster Children's Hospital (MCH)
* Diagnosed with PDA in need of treatment based on targeted neonatal echocardiography (TnEcho) performed prior to 27+6 CGA or postnatal age of 3 days, whichever comes later.
* Obtained parental consent.

Exclusion Criteria:

* Major congenital or genetic abnormalities
* Evidence for clinical or biochemical hepatic or renal failure (AST > 225 U/L, ALT > 150 U/L, or serum creatinine > 130 µmol/L)
* Sepsis - as defined by confirmed uncontrolled/active sepsis which will preclude any treatment of PDA
* Contraindications to receive oral ibuprofen:
* Severe hyperbilirubinemia in need for exchange transfusion
* Severe feeding intolerance
* Necrotizing enterocolitis (NEC)
* Gastrointestinal perforation
* Active bleeding
* Severe thrombocytopenia (< 50× 109/L)

Max Age: 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Estimated)
Dates: Start 2024-07-04 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Recruitment Feasibility | From intial dose to 96 hours after.
  Feasibility will be assessed by the ability to randomize at least 15% of all eligible patients during the study period.
Timeliness of PK Sample Result Availability | From initial dose to 96 hours after
  Feasibility will be assessed by the ability to obtain results for at least 80% of pharmacokinetic (PK) samples within 4 hours of sample collection.
Timeliness of Top-up Dosing Data for Intervention Arm | From initial dose to 96 hours after
  Feasibility will be assessed by the ability to generate dosing data for top-up administration within 14 hours of the previous dose in at least 80% of subjects in the intervention arm.
Timely Completion of Daily Targeted Neonatal Echocardiogram (TnEcho) | From initial dose to 96 hours after
  Feasibility will be assessed by the ability to perform daily TnEcho within 4 to 8 hours prior to the next scheduled dose in at least 80% of subjects.
Timely TnEcho Scoring and Model-Informed Precision Dosing (MIPD) Recommendation | From initial dose to 96 hours after
  Feasibility will be assessed by the ability to score the TnEcho, assign responsiveness grouping, and provide the MIPD recommendation for the second and third doses of oral ibuprofen within 24 hours of the previous dose in at least 80% of subjects.

SECONDARY OUTCOMES:
Achievement of Target Trough Concentration and AUC (Intervention Arm Only) | From first dose to 72 hours
  This exploratory outcome will evaluate the proportion of participants in the intervention arm who reach the predefined target trough concentration, AUC₀-₂₄, and AUC₀-₇₂. Results will be summarized descriptively and compared within the intervention group.
Maximum Ibuprofen Concentration (Cmax) ≤80 µg/mL (Intervention Arm Only) | From first dose to 72 hours
  This outcome will assess the proportion of intervention-arm participants whose maximum ibuprofen concentration (Cmax) remains at or below the predefined limit of 80 µg/mL. Results will be described and compared to the predefined threshold.
Daily Ibuprofen Dose ≤40 mg/kg (Intervention Arm Only) | From first dose to 72 hours
  This outcome will evaluate the proportion of participants in the intervention arm whose daily ibuprofen dose does not exceed 40 mg/kg. The frequency of participants meeting this dosing threshold will be summarized descriptively.
Closure of the Patent Ductus Arteriosus (PDA) | From first dose to 14 days
  This outcome will assess the proportion of participants with echocardiographically confirmed closure of the PDA following treatment. Results will be summarized and compared across study groups.
Need for Repeat Pharmacotherapy | From first dose to 14 Days
  This outcome will evaluate the proportion of participants requiring a repeat course of pharmacologic PDA treatment within 14 days of completing the initial course. Findings will be reported descriptively.
Need for Surgical Ligation | From first dose to 14 Days
  This outcome will assess the proportion of participants who require surgical ligation of the PDA due to persistent patency or clinical deterioration. Results will be summarized for both study groups.
Treatment Interruption | From first dose to 14 Days
  This outcome will describe the proportion of participants whose ibuprofen treatment was interrupted prior to completion due to clinical or safety concerns. Outcomes will be compared descriptively.
Occurrence of Adverse Events | From first dose to 14 Days
  This outcome will describe the proportion of participants who experience at least one adverse event during the follow-up period. Events will be classified by severity and relatedness to the study drug, and summarized descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Samira Samiee-Zafarghandy, MD, FRCPC, Principal Investigator — McMaster University
Locations (1):
- McMaster Children's Hospital - Neonatal Intensive Care Unit, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
This is a pilot feasibility study with a small sample size, and there are no current plans for data sharing.

REFERENCES:
- [Background] McEneny-King A, Foster G, Iorio A, Edginton AN. Data Analysis Protocol for the Development and Evaluation of Population Pharmacokinetic Models for Incorporation Into the Web-Accessible Population Pharmacokinetic Service - Hemophilia (WAPPS-Hemo). JMIR Res Protoc. 2016 Dec 7;5(4):e232. doi: 10.2196/resprot.6559. PMID 27927609
- [Background] Euteneuer JC, Kamatkar S, Fukuda T, Vinks AA, Akinbi HT. Suggestions for Model-Informed Precision Dosing to Optimize Neonatal Drug Therapy. J Clin Pharmacol. 2019 Feb;59(2):168-176. doi: 10.1002/jcph.1315. Epub 2018 Sep 11. PMID 30204236
- [Background] Van Overmeire B, Touw D, Schepens PJ, Kearns GL, van den Anker JN. Ibuprofen pharmacokinetics in preterm infants with patent ductus arteriosus. Clin Pharmacol Ther. 2001 Oct;70(4):336-43. PMID 11673749
- [Background] Hirt D, Van Overmeire B, Treluyer JM, Langhendries JP, Marguglio A, Eisinger MJ, Schepens P, Urien S. An optimized ibuprofen dosing scheme for preterm neonates with patent ductus arteriosus, based on a population pharmacokinetic and pharmacodynamic study. Br J Clin Pharmacol. 2008 May;65(5):629-36. doi: 10.1111/j.1365-2125.2008.03118.x. Epub 2008 Feb 27. PMID 18307541
- [Background] Engbers AGJ, Voller S, Flint RB, Goulooze SC, de Klerk J, Krekels EHJ, van Dijk M, Willemsen SP, Reiss IKM, Knibbe CAJ, Simons SHP. The Effect of Ibuprofen Exposure and Patient Characteristics on the Closure of the Patent Ductus Arteriosus in Preterm Infants. Clin Pharmacol Ther. 2022 Aug;112(2):307-315. doi: 10.1002/cpt.2616. Epub 2022 May 6. PMID 35429165
- [Background] Barzilay B, Youngster I, Batash D, Keidar R, Baram S, Goldman M, Berkovitch M, Heyman E. Pharmacokinetics of oral ibuprofen for patent ductus arteriosus closure in preterm infants. Arch Dis Child Fetal Neonatal Ed. 2012 Mar;97(2):F116-9. doi: 10.1136/adc.2011.215160. Epub 2011 Aug 11. PMID 21840880
- [Background] Samiee-Zafarghandy S, van Donge T, Fusch G, Pfister M, Jacob G, Atkinson A, Rieder MJ, Smit C, Van Den Anker J. Novel strategy to personalise use of ibuprofen for closure of patent ductus arteriosus in preterm neonates. Arch Dis Child. 2022 Jan;107(1):86-91. doi: 10.1136/archdischild-2020-321381. Epub 2021 May 11. PMID 33975823
- [Background] Mitra S, Florez ID, Tamayo ME, Mbuagbaw L, Vanniyasingam T, Veroniki AA, Zea AM, Zhang Y, Sadeghirad B, Thabane L. Association of Placebo, Indomethacin, Ibuprofen, and Acetaminophen With Closure of Hemodynamically Significant Patent Ductus Arteriosus in Preterm Infants: A Systematic Review and Meta-analysis. JAMA. 2018 Mar 27;319(12):1221-1238. doi: 10.1001/jama.2018.1896. PMID 29584842